CLINICAL TRIAL: NCT07326826
Title: Abdominal Wall Hernia Repair With Implantation of an Allogeneic Non-vascularised Rectus Abdominis Fascial Graft: A Pilot Prospective Observational Study
Brief Title: Hernia Repair Using Rectus Fascia Allograft
Status: Not yet recruiting | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Jiri Fronek, Professor of Surgery, MD, PhD, Institute for Clinical and Experimental Medicine
Other Study IDs: 48494/25
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Wall Hernia
Keywords: hernia repair; fascia; transplant; abdominal wall reconstruction
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Allogeneic non-vascularized rectus abdominis fascial graft (NVRF) — Elective incisional or primary ventral hernia repair with implantation of an allogeneic, non-vascularized rectus abdominis fascial graft (NVRF) to bridge/reinforce the abdominal wall fascial defect. The graft is prepared and implanted according to institutional standard procedures for tissue allografts, no vascular anastomosis is performed.

SUMMARY:
Abdominal wall closure in highly complex patients is one of the most difficult tasks in abdominal surgery. Repeated laparotomies, enterocutaneous fistulas, loss of the fascial layer and contaminated operative fields may prevent safe fascial approximation, and closure under high tension can lead to serious complications such as abdominal compartment syndrome. These problems are frequently encountered after intestinal or multivisceral transplantation and are not uncommon after liver transplantation. While component separation, flap techniques and mesh reinforcement are available, standard approaches may be insufficient or inappropriate in extensive or contaminated defects, and synthetic mesh may be contraindicated due to infection risk.

An allogeneic non-vascularized rectus abdominis fascial graft (NVRF) offers a practical alternative for isolated fascial defects with preserved skin coverage. The technique is relatively simple, reproducible, and does not require vascular reconstruction, potentially filling a gap where synthetic mesh is unsuitable. However, current evidence is limited, heterogeneous and largely retrospective.

This pilot prospective observational study will assess the feasibility and outcomes of elective incisional or primary ventral hernia repair using NVRF in (1) solid organ transplant recipients and (2) highly selected patients with exhausted standard abdominal wall reconstruction options and contraindications to synthetic mesh. Key outcomes include 12-month hernia recurrence, 90-day surgical site infection, immunologic response measured by donor-specific anti-HLA antibodies, direct healthcare costs over 12 months, and patient-reported quality of life using the EuraHS-QoL questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Solid organ transplant recipients (liver, kidney, pancreas, heart, or combined transplantation) ≥ 6 months post-transplantation with a primary ventral or incisional hernia.
* Non-transplant patients with a complex abdominal wall defect not amenable to currently established reconstructive methods (e.g., mesh repair, flap transposition, component separation).
* ECOG performance status 0-2.
* Written informed consent.

Exclusion Criteria:

* ECOG performance status 3-4.
* Pregnancy.
* High-dose corticosteroid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) undergoing elective incisional or primary ventral hernia repair with implantation of an allogeneic non-vascularized rectus abdominis fascial graft (NVRF). Eligible participants include solid organ transplant recipients at least 6 months post-transplant (liver, kidney, pancreas, heart, or combined transplants) and highly selected non-transplant patients with complex abdominal wall fascial defects not amenable to standard reconstruction (e.g., mesh repair, flap transposition, component separation) or with contraindications to synthetic mesh. Participants must provide written informed consent and have ECOG performance status 0-2. Pregnant patients, patietns with performance status ECOG 3-4, and on high-dose corticosteroid therapy are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-10 (Estimated); Study Completion 2029-02-10 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence | 12 months after surgery
  Cumulative incidence of hernia recurrence after the index hernia repair with NVRF (clinical and/or imaging-confirmed recurrence as per routine follow-up).

SECONDARY OUTCOMES:
Surgical site infection (SSI) | Up to 90 days after surgery
  Cumulative incidence of SSI within 90 days after the index surgery (any SSI diagnosed and treated according to institutional practice).
Donor-specific anti-HLA antibodies (DSA) | Baseline (day of surgery), 3 months, and 12 months
  Presence at baseline, de novo development, and change at 3 months, and 12 months after surgery.
Direct healthcare costs (public health insurance reimbursements) | 12 months after surgery
  Direct reimbursements associated with the index hospitalization for surgery and subsequent follow-up care over 12 months related to the surgery.
Patient-reported quality of life assessed using the European Hernia Society Quality of Life Questionnaire (EuraHS-QoL) | Baseline, 1 month and 12 months after surgery
  European Hernia Society Quality of Life Questionnaire is a disease-specific instrument evaluating pain, restriction of activities, and cosmetic discomfort.
  The total score ranges from 0 to 90, with higher scores indicating worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Froněk, prof., MD, PhD, FRCS, Principal Investigator — Institute for Clinical and Experimental Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Van De Winkel N, Muylle E, Canovai E, Amin I, Butler A, Vianna R, Selvaggi G, Farinelli P, Gondolesi G, Loinaz C, Justo I, Vilca-Melendez H, Skogsberg Dahlgren U, Herlenius G, Shamsaeefar A, Nikoupour H, Dubois A, Miserez M, D'Hoore A, Venick R, Pirenne J, Ceulemans LJ. Long-term Outcome After Nonvascularized Rectus Fascia Transplantation in Solid Organ Transplantation: A Global Multicenter IIRTA Survey. Transplant Direct. 2025 Jul 24;11(8):e1839. doi: 10.1097/TXD.0000000000001839. eCollection 2025 Aug. PMID 40718051
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40718051/